CLINICAL TRIAL: NCT01804504
Title: Survey on Eating Out Behavior and Dietary Structure in Urban Chinese Citizens and the Effect of Nutrition Education
Brief Title: Nutrition Education on the Metabolic Syndrome of Subjects Who Are Frequently Eating Out
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Second Military Medical University (Other)
Responsible Party: Principal Investigator, Donglian Cai, Professor, Second Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5186272761903
Record Dates: First submitted 2013-02-25; First posted 2013-03-05 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Eating out of home; Nutrition education
MeSH Terms: conditions — Metabolic Syndrome | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Food Frequency Questionnaire(FFQ) and KAP Questionnaire will be carried out before and after the trial to evaluate changes in calorie and nutrients intake, dietary structure, and KAP scores.
  Physical examination and biochemical examination before and after the trial.
- Nutrition education (Experimental): FFQ and KAP Questionnaire will be carried out before and after the trial to evaluate changes in calorie and nutrients intake, dietary structure, and KAP scores.
  Physical examination and biochemical examination before and after the trial.
  Do nutrition education
  Interventions: Behavioral: Nutrition education

INTERVENTIONS:
Behavioral: Nutrition education — The intervention group will be sent out a series of education materials, be arranged to attend lectures(once a month), dietary guidance or nutrition consultation at regular intervals(once every 2 weeks).
  Arms: Nutrition education

SUMMARY:
The project is aimed at investigating the effect of nutrition education on knowledge, attitude and practice (KAP)of subjects who are frequently eating out, and the effect on metabolic parameters.

DETAILED DESCRIPTION:
The project is aimed at investigating the dietary structure and frequencies of eating out via a cross-sectional study, on the basis of which a randomized, parallel controlled trials is to be carried out.The purpose is to evaluate the effect on metabolic parameters.

Hypotheses to be tested:Nutrition education has the effect of improving the metabolic parameters of subjects who are frequently eating out.

ELIGIBILITY:
Inclusion Criteria:

* Shanghai urban citizens
* Male or female 18 to 25 years of age;
* Frequently eat out(eat out 3 or more times per week);
* Clinical diagnosis of Metabolic Syndrome(Meet 3 or more Diagnostic criteria); A. Abdominal obesity: waist circumference>90cm ( M ), and>85cm( F ); B. Dyslipidemia:triglyceride≥1.7mmol/L; C. HDL-C < 1.04mmol/L; D. hypertension: blood pressure≥ 130/85mm Hg ( or have been diagnosed hypertension); E. Hyperglycemia : FPG≥6.1mmol/L and ( or ) 2-hour postprandial blood glucose≥7.8mmol/L and ( or ) have been diagnosed with diabetes;
* Signed written informed consent ;
* Can attend lectures.

Exclusion Criteria:

* Pregnant woman;
* Temporary resident population;
* Participating in another clinical trial 6 months before randomization.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Change in Body Weight | Baseline and 24 weeks
  Weight was obtained in light clothing to the nearest 0.1kg using a digital scale 8:00am and 10:00am after an overnight fast between.

SECONDARY OUTCOMES:
Change in Blood pressure | Baseline and 24 weeks
Change in waist circumference, waist hip ratio, waist to height | Baseline and 24 weeks
  Waist, hip circumference and height was measured using a plastic tape to the nearest 0.1 cm
Change in Waist, abdominal and hip circumference was measured using a plastic tape to the nearest 0.1 cm Change in fasting blood glucose | Baseline and 24 weeks
Change in serum triglyceride, cholesterol, HDL, LDL | Baseline and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Donglian Cai, Master, Principal Investigator — Shanghai Changhai Hospital ,Second Military Medical University
Locations (1):
- Changhai Hospital,Second Military Medical University, Shanghai, Shanghai Municipality, China